CLINICAL TRIAL: NCT04362774
Title: A Prospective, Multicenter, Open-label, Post-approval Study of the Safety and Effectiveness of ORBERA365 As a 12-month Adjunct to Weight Reduction for Obese Adults or Pre-surgical Weight Reduction for Obese or Super-obese Adults
Brief Title: ORBERA365 Post-Marketing Clinical Follow-up Study
Status: Terminated | Type: Observational
Why Stopped: Study was stopped after 1 site completed follow-up of enrolled patients, no other sites were opened in the study.
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTiMA365
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Overweight
Keywords: ORBERA
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: ORBERA365 — Behavioral modification program in conjunction with endoscopic placement of a single ORBERA365 Intragastric Balloon, filled with saline to an inflation volume between 400cc and 700cc with 2mL of Methylene blue (10mg/mL)

SUMMARY:
A prospective, multicenter, open-label, post-approval study of the safety and effectiveness of ORBERA36 as a 12-month adjunct to weight reduction for obese adults (BMI ≥ 27 kg/m2 and BMI ≤ 50 kg/m2) or for pre-surgical weight reduction in obese and super-obese adults (BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities).

DETAILED DESCRIPTION:
This is a prospective, multicenter, open label study of the safety and effectiveness of ORBERA365™ for use as an adjunct to behavioral modification for obese adults (BMI ≥ 27 kg/m2 and BMI ≤ 50 kg/m2) or for pre-surgical weight reduction in obese and super-obese adults (BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities). All study subjects will participate in a behavioral modification program for 52 weeks, which will include a low calorie diet as well as nutritional and behavior modification counseling. Subjects will have ORBERA365™ placed for up to 52 weeks.

Evaluations while on treatment will be performed at baseline (pre-placement), Day 0 (ORBERA365 placement) and during monthly clinic visits during the 1st 6 months of device therapy and at months 9 and ORBERA365 removal. All subjects will have a final study visit at 12 months, or study exit, whichever comes first. Device removal will occur at 52 unless removed early by subject request and/or physician recommendation. Reasons for early removal may include, but are not limited to, adverse events, subject dissatisfaction or achievement of weight loss goal.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult subjects;
2. BMI ≥ 27 kg/m2 and ≤ 50 kg/m2 if treatment is for temporary use for weight loss in subjects who failed to achieve and maintain weight loss with a supervised weight-control program;
3. BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities, if treatment is for pre-surgical temporary use for weight loss in order to reduce surgical risk
4. Be willing to commit to a long-term supervised diet and behavior modification program designed to increase the possibility of long-term weight loss maintenance;
5. Be able to follow the requirements outlined in the protocol, including complying with the visit schedule;
6. Be able to provide written informed consent;

Exclusion Criteria:

1. Presence of more than one ORBERA365 System Balloon at the same time;
2. Prior surgery of the esophagus, stomach, or duodenum;
3. Has any inflammatory disease of the gastrointestinal (GI) tract including esophagitis, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease;
4. Has any upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the GI tract such as atresias or stenosis;
5. Has a large hiatal hernia or hernia > 5 cm;
6. Has a structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the delivery catheter and/or an endoscope;
7. Has any other medical condition which would not permit elective endoscopy, such as poor general health or history and/or symptoms of severe renal, hepatic, cardiac, and/or pulmonary disease;
8. Has serious or uncontrolled psychiatric illness or disorder that could compromise subject understanding of or compliance with follow-up visits and removal of the device;
9. Alcoholism or drug addiction;
10. Unwilling to participate in an established medically-supervised diet and behavior modification program, with routine medical follow-up;
11. Taking a daily dose of aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants routinely and not under medical supervision;
12. Females who are pregnant, nursing, or planning a pregnancy within the next year;
13. Known to have, or suspected, allergy to materials contained in ORBERA365;
14. Participation in previous (within 60 days of study day 1) or ongoing clinical trial or current or past usage (within 60 days of study day 1) of investigational drug or device, or any use of an intragastric balloon prior to this study;
15. Genetically caused obesity;
16. Prior intragastric balloon therapy, bariatric surgery or considering bariatric surgery during the study;
17. Has a condition or is in a situation which in the Investigator's opinion may put the subject at significant risk or may interfere significantly with the subject's participation in the study.
18. Known gastrointestinal motility disorders, especially known delayed gastric emptying
19. Chronic use of anticholinergic medications and psychotropic medications known to delay gastric emptying.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adults who had already consented to receive ORBERA365 and who meet the eligibility criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Early Removal Percent | 12 months
  To demonstrate that the percentage of early removals for safety reasons (no including patient requests for removal related to achieving desired weight loss or inability to lose weight and have another procedure) is < 17.5%

SECONDARY OUTCOMES:
Total Body Weight Loss (%TBWL) Responders | 12 months
  To demonstrate >= 50% of completers will achieve >= 10% mean %TBWL at time of device removal. Completer is defined as maintaining device therapy for 12 months or successfully achieving weight loss goal (e.g. at least 5% TBWL) prior to device removal.
Adverse Events (AEs) | 12 months
  To assess the safety of ORBERA365 by summarizing the number of subjects with device- and procedure-related AEs.
% Total Body Weight Loss (%TBWL) | 12 months
  To estimate the %TBWL at 6, 9 and 12 months
% Excess Weight Loss (%EWL) | 12 months
  To estimate the %EWL at 6, 9, and 12 months, assuming an ideal weight based on having a BMI of 25 kg/m2
Body Mass Index (BMI) | 12 months
  To estimate the change from baseline in BMI at 9, 9 and 12 months.
Co-Morbidity Changes | 12 month
  To assess changes in obesity-related co-morbidities at 6, 9, and 12 months, if present at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Naveira, Study Director — Apollo Endosurgery, Inc.
Locations (1):
- Obymed, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
Only one investigator in this study